CLINICAL TRIAL: NCT01277185
Title: Calcium Metabolism in Mexican American Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Berdine Martin, Research Scientist, Nutrition Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Camp Calcium 11; 1R01HD061908-01A2 (NIH)
Record Dates: First submitted 2011-01-12; First posted 2011-01-14 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Osteoporosis
Keywords: calcium; healthy; Mexican-American adolescents; camp; girls; boys; bone
MeSH Terms: conditions — Osteoporosis; Muscle Cramp

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Calcium Diet (600-1200 mg/d) (Active Comparator)
  Interventions: Dietary Supplement: Low Calcium Diet
- High Calcium Diet (1100-2300mg/d) (Active Comparator)
  Interventions: Dietary Supplement: High Calcium Diet

INTERVENTIONS:
Dietary Supplement: Low Calcium Diet — The basal diet will contain 600 mg of Ca per day and constant sufficient amounts of all other nutrients. Additional Ca will be given unfortified beverages served three times per day. Teens will be randomized to a lower (600-1200 mg/d)level of calcium in the first camp followed by the opposite (higher calcium diet)regime in the second camp.
  Arms: Low Calcium Diet (600-1200 mg/d)
Dietary Supplement: High Calcium Diet — The basal diet will contain 600 mg of Ca per day and constant sufficient amounts of all other nutrients. Additional Ca will be given unfortified beverages served three times per day. Teens will be randomized to a higher (1100-2300mg/d)level of calcium in the first camp followed by the opposite (lower calcium diet)regime in the second camp.
  Arms: High Calcium Diet (1100-2300mg/d)

SUMMARY:
The purpose of this study is to identify calcium metabolism characteristics in Mexican American adolescents. The investigators predict that calcium requirements to maximize bone health in this population will be lower than for white youth but higher than their current intakes.

DETAILED DESCRIPTION:
Previously significant racial and sex differences in calcium retention and kinetics in adolescents has been found. Other minority groups have increased calcium absorption efficiency at low calcium intakes in contrast to white adolescents. Since Hispanics and specifically Mexican Americans will soon comprise an increasing proportion of our population. We propose to identify calcium metabolism characteristics in this group. We predict that calcium requirements to maximize bone health in this population will be lower than for white youth but higher than their current intakes.

Thus the specific aims of this project include:

* to establish calcium requirements
* to establish the relationship between calcium intake and calcium absorption
* to identify the major physiological parameters(kidney, intestine, bone) that contribute to calcium retention in Mexican-American adolescents

During this two-phase metabolic camp participants will consume either a higher calcium diet(1100-2300mg/d) or a lower calcium diet (600-1200mg/d) during the first 3-week phase and switch to the opposite regime during the second 3-week phase, with a 2-week washout period in between. Subjects will collect all excreta during both phases. Calcium absorption, height, weight, and bone density will evaluated throughout the 6-week period of the study.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy adolescents of Mexican American descent
* Mexican American boys age 13-15
* Mexican American girls age 12-14

Exclusion Criteria:

* Malabsorptive disorders
* Anemia
* Smoking
* History of medications known to affect calcium metabolism
* Body weight outside 85-120% of ideal body weight for height
* Regular consumption of illegal drugs
* Contraceptive use
* Pregnancy

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2010-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Calcium Absorption and Retention | June 2010-July 2010

SECONDARY OUTCOMES:
Bone Density | June 2010-July 2010

CONTACTS AND LOCATIONS:
Overall Officials: Connie Weaver, PhD, Principal Investigator — Purdue University; Berdine Martin, PhD, Study Director — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Palacios C, Martin BR, McCabe GP, McCabe L, Peacock M, Weaver CM. Dietary calcium requirements do not differ between Mexican-American boys and girls. J Nutr. 2014 Aug;144(8):1167-73. doi: 10.3945/jn.113.188318. Epub 2014 May 28. PMID 24872223